CLINICAL TRIAL: NCT01235988
Title: Systematic Review of the Clinical and Cost Effectiveness of Treatments for Idiopathic (Immune) Thrombocytopenic Purpura (ITP): Direct Meta Analysis
Brief Title: Meta-analysis - Eltrombopag
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114013
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Thrombocytopaenia
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eltrombopag & standard of care
  Interventions: Drug: Eltrombopag
- Standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag 50mg & standard of care
  Groups: Eltrombopag & standard of care
Drug: Placebo — Placebo + standard of care
  Groups: Standard of care

SUMMARY:
The purpose of the meta-analysis was to explore the efficacy of eltrombopag versus placebo (standard of care)

DETAILED DESCRIPTION:
Meta-analysis of three studies: Bussell 2007 & Bussell 2009 & RAISE (TRA102537).

ELIGIBILITY:
Inclusion Criteria:

* Adults with ITP
* Received a pre-specified treatment
* Prospective clinical studies with at least 10 patients

Exclusion Criteria:

* Subjects with ITP due to other causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meta-analysis: A systematic review was conducted to obtain all relevant evidence relating to eltrombopag and relevant studies were selected
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
>=50 Gi/L platelet count to <400 Gi/L | 43 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline